CLINICAL TRIAL: NCT07218562
Title: PATH to Reducing Burnout Among Peers Who Deliver Harm Reduction Services: Improving Workforce and Service System Outcomes Through a Combined eLearning and Group Consultation Intervention (R61 Phase Pilot)
Brief Title: PATH (Peer Advanced Training in Harm Reduction) to Reducing Burnout Among Peers Who Deliver Harm Reduction Services (R61 Phase Pilot)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dennis Watson, Senior Research Scientist, Chestnut Health Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R61DA061340 (NIH)
Record Dates: First submitted 2025-09-30; First posted 2025-10-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Burnout; Compassion Satisfaction; Secondary Trauma
Keywords: peer recovery support specialist; harm reduction training; opioid use disorder; substance use disorder
MeSH Terms: conditions — Burnout, Psychological; Compassion Fatigue; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATH pilot participants (Experimental): Receive PATH pilot intervention
  Interventions: Behavioral: PATH (Peer Advanced Training in Harm reduction)

INTERVENTIONS:
Behavioral: PATH (Peer Advanced Training in Harm reduction) — PATH is an educational workforce intervention for improving peer recovery support specialists' (PRSS) harm reduction (HR) service delivery ability and quality and as a PRSS workforce and service system support. PATH will include 3 hours of eLearning modules and 8 weekly ECHO (Extension for Community Health Outcomes) meetings lasting 1.5 hours each, delivered over 2 months. Each ECHO session includes a 30-minute presentation followed by one hour of case-based discussion about a real client or problem. The entire PATH intervention will take 15 hours (3 hours of eLearning and 12 hours of ECHO participation) over 3 months. Participants are expected to complete all 15 hours, completing the 3 hours of eLearning before starting the 12 hours of ECHO activities.

SUMMARY:
The investigators propose to develop and test the effectiveness of PATH (Peer Advanced Training in Harm reduction) as an educational workforce intervention for improving peer recovery support specialists' (PRSS) harm reduction (HR) service delivery ability and quality and as a PRSS workforce and service system support. The PATH intervention combines (a) virtual education and (b) case-based consultation. The investigators hypothesize that PATH will improve organizational-level PRSS burnout, additional workforce outcomes, and HR service quality.

DETAILED DESCRIPTION:
The investigators will pilot the PATH intervention with two Recovery Community Organizations (RCOs) to understand its acceptability, appropriateness, and feasibility. Administrator(s)/supervisor(s) will participate in PATH alongside their peer recovery support specialist (PRSS) staff.

PATH will include 3 hours of eLearning modules and 8 weekly ECHO (Extension for Community Health Outcomes) meetings lasting 1.5 hours each, delivered over 2 months. Each ECHO session includes a 30-minute presentation followed by one hour of case-based discussion about a real client or problem. The full PATH intervention will take 15 hours (3 hours of eLearning and 12 hours of ECHO participation) over 3 months. Participants are expected to complete all 15 hours, completing the 3 hours of eLearning before starting the 12 hours of ECHO activities.

The investigators will administer the PATH components with the PRSS and administrators/supervisors from two RCOs, while assessing the duration and dose of an individual participant's engagement by tracking eLearning module completion and ECHO attendance. Voluntary survey and qualitative data collection will be used to assess the primary measures for this pilot. Data collection will also assess training satisfaction and changes in burnout, compassion satisfaction, secondary trauma, and HR knowledge, attitudes, and skills.

Participants of the PATH pilot will be invited to complete surveys at three timepoints. The baseline survey will be distributed immediately prior to beginning the PATH training activities. Measures on the baseline survey will include demographics, burnout, compassion satisfaction, secondary trauma, and HR knowledge, attitudes, and skills. Following the completion of the eLearning components of the training (approximately 1 month post-initiation), the second survey will be distributed to all participants. Measures on the survey will include acceptability, appropriateness, and feasibility of the training component, as well as training satisfaction. Finally, following completion of the final ECHO meeting (approximately 3 months post-initiation), the third survey will be distributed to all participants. All measures from the first two surveys will be included in the final survey, excluding demographics. All surveys will be collected in REDCap. Personalized survey links will be sent directly to each participant's email address. Each survey will take approximately 15-30 minutes to complete. Additionally, the investigators will track and obtain administrative training data for the eLearning modules and ECHO meetings, including engagement and attendance.

PRSS staff participants will also be invited to complete a final qualitative focus group regarding their participation in the PATH training activities. Depending on the final number of participants per RCO, investigators will conduct 1-2 focus groups for each site. Each focus group will last approximately 60-90 minutes and be conducted via Zoom teleconference. Questions will focus on participants' experiences with the PATH training activities, particularly regarding the content, clarity, applicability, relevance, and usefulness of both the eLearning modules and ECHO meetings. Additionally, participants will be asked about barriers and facilitators to completing the PATH training activities and suggestions for improvement. Similarly, the administrator/supervisor will be invited to complete a final qualitative interview regarding their organization's participation in the PATH training activities. The interview will last approximately 45-60 minutes and be conducted via Zoom teleconference. Questions will focus on the administrator's opinions of staff experiences with the PATH training activities, particularly regarding the applicability, relevance, and usefulness of both the eLearning modules and ECHO meetings, as well as the impact of the training on their team. Administrators/supervisors will be asked about barriers and facilitators to having their staff complete the PATH training activities and suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

* employed at a Recovery Community Organization or an organization providing direct harm reduction services, including syringe and/or outreach services
* current PRSS staff or administrator involved in HR service delivery
* is at least 18 years of age.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability, Appropriateness, and Feasibility | Baseline - 3 months
  Measured using the Acceptability, Appropriateness, and Feasibility Scales (AIM, IAM, FIM), a brief validated 4-item instruments measuring participants' perceptions of the intervention's relevance, practicality, and fit for their work.
Training Satisfaction | Baseline - 3 Months
  Measured using the Training Satisfaction Questionnaire, a custom Likert-scale survey assessing overall satisfaction with the learning experience, content relevance, and applicability to peer support practice.

OTHER OUTCOMES:
Burnout | Baseline - 3 months
  Measures mean PRSS Burnout using the 10-item burnout subscale from the Professional Quality of Life (ProQOL) scale. Questions ask respondents to rate how often they have experienced items listed in their work over the past 30 days on a 5-point Likert scale (1/"Never"-5/"Very often").
Compassion satisfaction and secondary traumatic stress | Baseline - 3 months
  Measured using the 10-question Compassion Satisfaction and Secondary Traumatic Stress job sub-scales from the Professional Quality of Life Scale (v.5). Questions ask respondents to rate how often they have experienced items listed in their work over the past 30 days on a 5-point Likert scale (1/"Never"-5/"Very often").
Harm-Reduction Knowledge, Attitudes, and Skills | Baseline - 3 months
  Measured using the Harm-Reduction Knowledge, Attitudes, and Skills (HR-KAS), a 13-item custom scale assessing conceptual understanding and application of harm-reduction principles in peer recovery work. Participants are asked to rate each item on a 10-point Likert scale. Sub scale includes: knowledge (4 items; 1/no knowledge-10/high level of knowledge), attitudes (4 items; 1/strongly disagree-10/strongly agree), skills (5 items; 1/cannot do at all-10/highly certain). Six original questions (1 knowledge, 2 attitude, and 3 skill questions) specific to this study have been added.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Watson, PhD, Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems Lighthouse Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual and aggregate PRSS survey data (raw and recoded) will be shared publicly after completing all data and analyses. Files will be shared in the format most relevant to the software used to develop them, as well as CSV files.
  De-identified qualitative transcripts will be maintained and shared only with an established data-sharing agreement. Files containing coding lists and summaries and transcript attributes will also be shared with appropriate agreements in place. Open sharing of qualitative data may risk identifying participants, particularly in small rural organizations where contextual details are difficult to mask. Standard protections, like de-identification and Certificates of Confidentiality, may be insufficient.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: The study protocol, statistical analysis plan, and informed consent form will be made publicly available on Open Science Framework.